CLINICAL TRIAL: NCT07276620
Title: A Study on the Efficacy and Safety of Ivarmacitinib in the Treatment of Moderate to Severe Atopic Dermatitis in Adolescents and Adults
Brief Title: Treatment of Moderate-to-Severe Atopic Dermatitis With Ivarmacitinib in Adolescents and Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-DER-RWS-101
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis; Ivarmacitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Moderate-to-Severe Atopic Dermatitis with Ivarmacitinib in Adolescents and Adults (Experimental)
  Interventions: Drug: Ivarmacitinib Sulfate Tablets

INTERVENTIONS:
Drug: Ivarmacitinib Sulfate Tablets — Patients with moderate to severe atopic dermatitis are initially treated with 4 mg of ivarmacitinib once daily for 16 weeks. Subsequently, those who respond adequately may transition to an individualized maintenance regimen until week 52.If a suboptimal response is observed with the 4 mg once-daily dose, an increase to 8 mg once daily may be considered. Treatment should be discontinued if an adequate response is not achieved following dose escalation to 8 mg once daily.

SUMMARY:
Atopic dermatitis (AD) is a skin condition characterized by a rash and itching, resulting from skin inflammation. Ivarmacitinib is an approved medication for treating AD.

This study aims to evaluate the effectiveness and safety of Ivarmacitinib in the treatment of moderate-to-severe atopic dermatitis under real-world conditions. It will assess the time to pruritus improvement and skin lesion clearance, collect large-sample safety data, analyze disease improvement across patient subgroups with different baseline characteristics, and explore the impact of various maintenance treatment regimens on disease recurrence.

It is expected that there will be no additional burden for participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 75 years;
* Diagnosed with moderate-to-severe atopic dermatitis (AD) ;
* Participants (and legal representatives for adolescents) able to understand and communicate with the investigator.

Exclusion Criteria:

* Subject has any of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

  1. Absolute lymphocyte count of <0.50 x 10^9 /L (<500/mm3);
  2. Absolute Neutrophil Count (ANC) of <1 X 10^9/L (<1000/mm3);
  3. Hemoglobin level < 80 g/L.
* Subject has any malignancies or has a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Subject with a prior history of thromboembolic events, including deep vein thromboses (DVT), pulmonary embolism, cerebrovascular accidents and those with known inherited conditions that predispose to hypercoagulability.
* Presence of an active severe acute or chronic bacterial, fungal, or viral infection requiring systemic therapy.
* Subjects with active tuberculosis or known active hepatitis B and/or hepatitis C infection.
* Subjects with clinically significant diseases of the heart, liver, kidney, or other major organ systems.
* Female subject who is pregnant, breastfeeding, or considering pregnancy during the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving at Least a 75% Reduction in Eczema Area and Severity Index Score (EASI 75) From Baseline at Week 16 | Baseline and Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic dermatitis based on assessments of the head/ neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness , thickness, scratching, and lichenification.
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.

SECONDARY OUTCOMES:
Time to achieve a ≥4-point improvement from baseline in the Worst Itch Numerical Rating Scale (WI-NRS). | Baseline and Day 7
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
The proportion of patients achieving an Investigator's Global Assessment (IGA) response at each scheduled visit, defined as an IGA score of 0 or 1 with at least a 2-point reduction from baseline. | Baseline and Week 1、2、4、8、12、16、24、32、40、52
  The IGA is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  0 - Clear: No inflammatory signs of AD;
  1. - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification, no oozing or crusting;
  2. - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification, no oozing or crusting;
  3. - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  4. - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
The proportion of subjects achieving EASI 75 at each scheduled visit. | Baseline and Week 1、2、4、8、12、24、32、40、52
Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Patient Oriented Eczema Measure (POEM) Total Score | Baseline and Week 1、2、4、8、12、16、24、32、40、52
  The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults.
  Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). A change in POEM score of 3.4 points is considered the minimal clinically important difference.
Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Dermatology Life Quality Index (DLQI) | Baseline and Week 1、2、4、8、12、16、24、32、40、52
  The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
The recurrence of atopic dermatitis. | Week 16、52
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From Baseline to 30 days following last dose of study drug (Week 52)